CLINICAL TRIAL: NCT04182529
Title: Photo Neuro-Modulation Therapy to Middle Aged and Older Adults With Mild Memory Problem
Brief Title: Photo Neuro-Modulation Therapy to Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Chan Sui-yin Agnes, Professor Chan Sui-yin Agnes, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017.354
Record Dates: First submitted 2019-11-22; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Photo Neuro-Modulation Therapy, Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photoneuromodulation Therapy (Experimental): In this study low-level LED near-infrared (670-810nm) including MedX Health Model 1100 or WiseFori5-3800 will be used. The United States Food and Drug Administration (FDA) has approved this type of device as imposing insignificant risk (FDA-cleared for home treatment, 2005). At each visit, LED clusters will be applied simultaneously for 20 minutes on the Fp1, Fp2 and Pz regions according to the International 10-20 system (Homan, Herman and Purdy, 1987) (energy density, 13 Joules/cm2 [J/cm2] per each LED cluster head placement). The total LED treatment time per visit was 20 minutes.
  Interventions: Device: Photoneuromodulation therapy
- Control Group (Sham Comparator): Subject will not be given any active stimulation
  Interventions: Other: Sham

INTERVENTIONS:
Device: Photoneuromodulation therapy — low-level LED near-infrared (670-810nm) including MedX Health Model 1100 or WiseFori5-3800
  Arms: Photoneuromodulation Therapy
Other: Sham — Sham, no active stimulation will be given to subjects
  Arms: Control Group

SUMMARY:
It is well-documented that mild cognitive impairment (MCI) is associated frontal lobe dysfunction and executive dysfunction. In addition, many studies reported high level of MCI symptoms among the elderly and the trend is increasing in Hong Kong. Based upon the link between MCI and frontal and executive function problems, it is conceivable that elderly who exhibits high levels of memory problems would exhibit frontal and executive function problems. To our knowledge, there is still a lack of effective treatment or therapy for MCI, it is important to investigate effective intervention that can efficiently improve the cognitive ability of MCI patients or patients with mild memory problems. The objective of the present study is to compare individuals with mild memory problems after the Photo neuro-modulation Therapy (PNMT) and those who do not. 40 middle aged and older adults were recruited from the subject database of the Neuropsychology Laboratory of The Chinese University of Hong Kong. Participants were divided randomly and equally into treatment group, as well as the placebo group. Several computerized executive function tests will be used before and after the treatment under the recording of near-infrared spectroscopy (NIRS), which estimates level of frontal activation. It is hypothesized that compared to participants without PNMT, those with PNMT will have a better performance in the executive function tasks and exhibit a higher frontal activation. The cognitive and neurophysiological results would provide evidences on the possibility of PNMT in treating individuals with mild memory problems, as well as with other mental disorders.

ELIGIBILITY:
Inclusion Criteria:

* 40 middle age and older adults with aged 40 or above who have subjective memory complaints

Exclusion Criteria:

* A history of head injury, or any neurological/psychiatric disorders, and dementia will be excluded. In addition, a score higher than 7 on the short form of the Chinese Geriatric Depression Scale (CGDS-SF; Lee, Chiu, Kwok, & Leung, 1993)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
N-Back Test (cognitive test battery) | through study completion, an average of 2 year
  a digit n-back paradigm to assess working memory
Category Fluency Test | through study completion, an average of 2 year
  a test to assess the ability to generate words that belong to a semantic category in a controlled manner
The Hong Kong List Learning Test | through study completion, an average of 2 year
  a tests to assess memory function of the participants
The Chinese Version of the Mattis Dementia Rating Scale | through study completion, an average of 2 year
  a test to estimate the global functioning level of the participants, lowest score is 0, highest score is 144, higher score means better global functioning level
NIRS Recording | through study completion, an average of 2 year
  NIRS to record the hemodynamic response, measured in mmol/mm
EEG Recordings | through study completion, an average of 2 year
  EEG is used to record electrical activity of the brain, measured in microvolts, EEG power spectrum
EEG Recordings | through study completion, an average of 2 year
  EEG source localisation, measured in current density

CONTACTS AND LOCATIONS:
Locations (1):
- Neuropsychology Laboratory, Department of Psychology, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided